CLINICAL TRIAL: NCT00065013
Title: Strength Training Following Gastric Bypass for Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Allan Geliebter, St. Luke's-Roosevelt Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: STGASB (completed); R03DK061519 (NIH)
Record Dates: First submitted 2003-07-16; First posted 2003-07-18 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2010-01

CONDITIONS: Obesity
Keywords: obesity; gastric bypass; obesity surgery; bariatric surgery; exercise
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: strength training

SUMMARY:
We will assess whether undesirable loss of lean tissue following gastric bypass surgery for obesity can be minimized by protein supplementation and exercise training.

ELIGIBILITY:
* clinically severe obesity
* candidate for bypass surgery
* new york city local address
* willing to visit hospital weekly

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2003-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Geliebter, PhD, Principal Investigator — St. Luke's-Roosevelt Hospital Center

REFERENCES:
- See also: Related Info — http://www.nyorc.org/